CLINICAL TRIAL: NCT04145258
Title: Intensified Tuberculosis Treatment to Reduce the Mortality of HIV-infected and Uninfected Patients With Tuberculosis Meningitis: a Phase III Randomized Controlled Trial (Acronym: INTENSE-TBM)
Brief Title: Intensified Tuberculosis Treatment to Reduce the Mortality of Patients With Tuberculous Meningitis
Acronym: INTENSE-TBM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: European Union (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANRS 12398 INTENSE-TBM; EDCTP RIA2017T-2019 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2019-10-22; First posted 2019-10-30 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Tuberculous Meningitis
Keywords: Tuberculous Meningitis; Intensified treatment; High dose Rifampicin; Linezolid; Aspirin; Subsaharan Africa
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be open-label for anti-TB treatment and placebo-controlled for aspirin treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WHO TBM treatment + placebo (Other): * Inclusion (D-0) to end of Week-8 (W-8): isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d + ethambutol 20 mg/kg/d + pyrazinamide 30 mg/kg/d + placebo of aspirin
  * W-9 to W-40: isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d.
  Interventions: Drug: Placebo of aspirin; Drug: WHO TBM treatment
- WHO TBM treatment + aspirin (Other): * Inclusion (D-0) to end of Week-8 (W-8): isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d + ethambutol 20 mg/kg/d + pyrazinamide 30 mg/kg/d + aspirin 200 mg/d
  * W-9 to W-40: isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d.
  Interventions: Drug: Aspirin; Drug: WHO TBM treatment
- Intensified TBM treatment + placebo (Other): * Inclusion (D-0) to end of Week-8 (W-8): high dose rifampicin (35 mg/kg/d) + high dose linezolid (1200 mg/d from D-0 to end of W-4, then 600 mg/d from W-5 to W-8) + isoniazid 5 mg/kg/d + ethambutol 20 mg/kg/d + pyrazinamide 30 mg/kg/d + placebo of aspirin
  * W-9 to W-40: isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d.
  Interventions: Drug: Placebo of aspirin; Drug: Intensified TBM treatment
- Intensified TBM treatment + aspirin (Other): * Inclusion (D-0) to end of Week-8 (W-8): high dose rifampicin (35 mg/kg/d) + high dose linezolid (1200 mg/d from D-0 to end of W-4, then 600 mg/d from W-5 to W-8) + isoniazid 5 mg/kg/d + ethambutol 20 mg/kg/d + pyrazinamide 30 mg/kg/d + aspirin 200 mg/d
  * W-9 to W-40: isoniazid 5 mg/kg/d + rifampicin 10 mg/kg/d.
  Interventions: Drug: Aspirin; Drug: Intensified TBM treatment

INTERVENTIONS:
Drug: Aspirin — Two tablets of aspirin 100 mg per day from inclusion (D-0) to end of Week-8 (W-8)
  Arms: Intensified TBM treatment + aspirin; WHO TBM treatment + aspirin
Drug: Placebo of aspirin — Two placebo tablets with the same appearance of aspirin 100 mg per day from inclusion (D-0) to end of Week-8 (W-8)
  Arms: Intensified TBM treatment + placebo; WHO TBM treatment + placebo
Drug: WHO TBM treatment — 2 months of (R-H-Z-E) + 7 months of (R-H)
  Other Names: Standard WHO treatment for TB meningitis
  Arms: WHO TBM treatment + aspirin; WHO TBM treatment + placebo
Drug: Intensified TBM treatment — 2 months of (HDR-L-H-Z-E) + 7 months of (R-H), with HDR=high-dose rifampicin and L=linezolid
  Arms: Intensified TBM treatment + aspirin; Intensified TBM treatment + placebo

SUMMARY:
INTENSE-TBM is randomized controlled, phase III, multicenter, 2 x 2 factorial plan superiority trial assessing the efficacity of two interventions to reduce mortality from tuberculous meningitis (TBM) in adolescents and adults with or without HIV-infection in sub-Saharan Africa:

* Intensified TBM treatment with high-dose rifampicin and linezolid, compared to WHO standard TBM treatment.
* Aspirin, compared to not receiving aspirin. The trial will be open-label for anti-TB treatment and placebo-controlled for aspirin treatment.

DETAILED DESCRIPTION:
Settings: Côte d'Ivoire, Madagascar, Uganda, South Africa.

Follow-up: Participants will be followed up for 40 weeks.

Sample size: 768 patients (192 in each arm).

Primary analysis: We will use a Cox proportional hazard ratio model to compare intensified TB treatment with WHO standard TB treatment, and aspirin with placebo, adjusting for the initial stratification variables (trial country, HIV status, British Medical Research Council |BMRC] severity grade). The primary analysis will be conducted in the intention to treat population.

Sub-studies:

* The PK-PD sub-study will take place in the 4 participating countries, and involve 40 participants in total.
* The Multi-Omics sub-study will only take place in South-Africa. It will involve 160 participants in this country.

Participants in each sub-study will sign a specific informed consent.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 15 years
2. TBM defined as "definite", "probable" or "possible"
3. Signed Informed Consent

   * Definite TBM = at least one of the following criteria: acid-fast bacilli seen in CSF microscopy, positive CSF M. tuberculosis culture, or positive CSF M. tuberculosis commercial nucleic acid amplification test.
   * Probable TBM = total modified Marais score ≥12 when neuroimaging is available, or ≥10 when neuroimaging is not available (at least 2 points should come from CSF or cerebral imaging criteria).
   * Possible TBM = total modified Marais 6-11 when neuroimaging is available, or 6-9 when neuroimaging is not available.

Exclusion criteria:

* > 5 days of TB treatment
* Renal failure (eGFR<30 ml/min, CKD-EPI formula).
* Neutrophil count < 0.6 x 109/L.
* Hemoglobin concentration < 8 g/dL.
* Total bilirubin > 2.6 times the Upper Limit of Normal
* Platelet count < 50 x 109/L.
* ALT > 5 times the Upper Limit of Normal.
* Clinical evidence of liver failure or decompensated cirrhosis.
* For women: more than 17 weeks pregnancy or breastfeeding.
* For patients without decrease level of consciousness (Glasgow Coma Scale = 15): Peripheral neuropathy scoring Grade 3 or above on the Brief Peripheral Neuropathy Score (BPNS).
* Documented M. tuberculosis resistance to rifampicin.
* Positive gram-stain, bacterial culture or cryptococcal antigen in the Cerebral Spinal Fluid.
* Evidence of active bleeding (hemoptysis, gastrointestinal bleeding, hematuria, intracranial bleeding).
* Inability to collect Cerebral Spinal Fluid, except for patients with confirmed tuberculosis (by rapid molecular test or culture) from another biological sample and clinical and/or CT scan evidence of meningitis.
* Major surgery within the last two weeks prior to inclusion.
* Ongoing chronic aspirin treatment (eg for cardiovascular risk).
* Current use of drugs contraindicated with study drugs and that cannot be safely stopped (see Appendix 1: Drugs contra-indicated with study drugs).
* In available history from patients:

  * Evidence of past intracranial bleeding.
  * Evidence of past of peptic ulceration.
  * Evidence of recent (< 3 month) gastrointestinal bleeding.
  * Known hypersensitivity contraindicating the use of study drugs .
  * Evidence of porphyria.
  * Evidence of hyperuricemia or gout.
* Any reason which at the discretion of the investigator would compromise safety and cooperation in the trial.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2021-02-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause death | Up to 40 weeks

SECONDARY OUTCOMES:
Rate of all-cause death | Up to 8 weeks
Rate of all-cause death or loss to follow-up | Up to 40 weeks
Rate of new central neurological event or aggravation of a central neurological event existing at baseline | Up to 40 weeks
Rate of grade 3-4 adverse events (DAIDS adverse events grading table) | Up to 40 weeks
Rate of serious adverse events | Up to 40 weeks
Rate of solicited treatment related adverse events | Up to 40 weeks
Percentage of patients with disability | 40 weeks
M. tuberculosis culture conversion rate | 1 week and 4 weeks
Time to culture positivity | Up to 40 weeks
Time to first hospital discharge | Up to 40 weeks
Cost-effectiveness incremental ratio of trial interventions | Up to 40 weeks
Prevalence of resistance to anti-TB drugs among patients with positive culture at inclusion | Up to 40 weeks
Subset of patients: In vitro bactericidal activity of anti-TBM treatment | 1 week and 4 weeks
Subset of patients: Maximum Plasma Concentration [Cmax] of rifampicin and linezolid | 1 week and 4 weeks
  Plasma Cmax, cerebrospinal fluid [CSF] Cmax, and plasma/CSF Cmax ratio
Subset of patients: Minimum Plasma Concentration [Cmin] of rifampicin and linezolid | 1 week and 4 weeks
  Plasma Cmin, cerebrospinal fluid [CSF] Cmin, and plasma/CSF Cmin ratio
Subset of patients: Area Under the Curve [AUC] of rifampicin and linezolid | 1 week and 4 weeks
  Plasma AUC, cerebrospinal fluid [CSF] AUC, and plasma/CSF AUC ratio
Subset of patients: Time for maximal concentration [Tmax] of rifampicin and linezolid | 1 week and 4 weeks
  Plasma Tmax, cerebrospinal fluid [CSF] Tmax, and plasma/CSF Tmax ratio
Subset of patients: Half-life (t1/2) of rifampicin and linezolid | 1 week and 4 weeks
  Plasma t1/2, cerebrospinal fluid [CSF] t1/2, and plasma/CSF t1/2 ratio
HIV-infected participants: Rate of new AIDS-defining illnesses | Up to 40 weeks
HIV-infected participants: Percentage of participants with virological success (plasma HIV-1 RNA <50 copies/ml) | 28 weeks and 40 weeks
HIV-infected participants: CD4 count change from baseline | 28 weeks and 40 weeks
HIV-infected participants, subset of patients: Maximum Plasma Concentration [Cmax] of of dolutegravir | 1 week and 4 weeks
  Plasma Cmax, cerebrospinal fluid [CSF] Cmax, and plasma/CSF Cmax ratio
HIV-infected participants, subset of patients: Minimum Plasma Concentration [Cmin] of dolutegravir | 1 week and 4 weeks
  Plasma Cmin, cerebrospinal fluid [CSF] Cmin, and plasma/CSF Cmin ratio
HIV-infected participants, subset of patients: Area Under the Curve [AUC] of dolutegravir | 1 week and 4 weeks
  Plasma AUC, cerebrospinal fluid [CSF] AUC, and plasma /CSF AUC ratio
HIV-infected participants, subset of patients: Time for maximal concentration [Tmax] of dolutegravir | 1 week and 4 weeks
  Plasma Tmax, cerebrospinal fluid [CSF] Tmax, and plasma /CSF Tmax ratio
HIV-infected participants, subset of patients: Half-life (t1/2) of dolutegravir | 1 week and 4 weeks
  Plasma t1/2, cerebrospinal fluid [CSF] t1/2, and plasma/CSF t1/2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bonnet, M.D., Ph.D., Principal Investigator — University Hospital, Bordeaux
Locations (13):
- Côte d’Ivoire (3):
  - Cocody University Hospital, Abidjan
  - Treichville University Hospital, Abidjan
  - Yopougon University Hospital, Abidjan
- Madagascar (3):
  - University Hospital Joseph Raseta Befelatanana, Antananarivo
  - University Hospital Tambohobe, Fianarantsoa
  - Morafeno University Hospital, Toamasina
- South Africa (5):
  - Kayelitsha District Hospital, Cape Town
  - Mitchells Plain Hospital, Cape Town
  - New Somerset Hospital, Cape Town
  - Dora Nginza Hospital, Port Elizabeth
  - Livingstone and PE Central Hospitals, Port Elizabeth
- Uganda (2):
  - Mbarara Regional Reference Hospital, Mbarara
  - Regional Reference Hospital of Kabale, Mbarara

REFERENCES:
- [Derived] Maitre T, Bonnet M, Calmy A, Raberahona M, Rakotoarivelo RA, Rakotosamimanana N, Ambrosioni J, Miro JM, Debeaudrap P, Muzoora C, Davis A, Meintjes G, Wasserman S, Wilkinson R, Eholie S, Nogbou FE, Calvo-Cortes MC, Chazallon C, Machault V, Anglaret X, Bonnet F. Intensified tuberculosis treatment to reduce the mortality of HIV-infected and uninfected patients with tuberculosis meningitis (INTENSE-TBM): study protocol for a phase III randomized controlled trial. Trials. 2022 Nov 8;23(1):928. doi: 10.1186/s13063-022-06772-1. PMID 36348453
- See also: INTENSE-TBM project website — https://intense-tbm.org/